CLINICAL TRIAL: NCT02273895
Title: Development of a Diagnostic Tool for Alzheimer's Disease
Brief Title: The Use of EEG in Alzheimer's Disease, With and Without Scopolamine - A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mentis Cura (Industry)
Collaborators: Landspitali University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MC-CT-001
Record Dates: First submitted 2014-09-29; First posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: AD
Keywords: Scopolamine, AD, EEG, MCI
MeSH Terms: interventions — Scopolamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Active Comparator): Scopolamine
  Interventions: Drug: Scopolamine
- MCI (Active Comparator): Scopolamine
  Interventions: Drug: Scopolamine
- AD (Active Comparator): Scopolamine
  Interventions: Drug: Scopolamine

INTERVENTIONS:
Drug: Scopolamine — 0.3 mg/mL, intravenously, once
  Other Names: Scopolamine hydrobromide

SUMMARY:
The objective of this study is to compare the electroencephalography (EEG) responses of three distinct groups of individuals to scopolamine: 1) a group of Alzheimer Dementia (AD) patients, 2) a group of individuals suffering from Mild Cognitive Impairment (MCI) and 3) a group of controls. The main purpose of this comparison is to discover ways to use these responses to distinguish between the group of AD patients and controls in order to develop a diagnostic tool for AD. The purpose of including the MCI group is to investigate whether this diagnostic tool can predict which member of the MCI group will develop AD later in life.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects:

* Between 60-80 years of age.
* Volunteers will have to be in good general health as determined by standard physical examination.
* Normal Electrocardiograph (ECG)

MCI subjects:

* Diagnosed with MCI at the Memory Clinic at the Landspitali University Hospital using F 06,7 according to International Classification of Diseases (ICD) - 10.
* Between 60-80 years of age.
* Subjects need to score between 2 and 3 on the Global Deterioration Scale (GDS).
* Normal ECG

Alzheimer's patients:

* Diagnosed with AD according to ICD - 10 in Follow up at the Memory Clinic at the Landspitali University Hospital.
* Between 60-80 years of age.
* Subjects need to score between 3-5 on the GDS.
* Normal ECG
* Treated with Reminyl® for the Alzheimer disease.

Exclusion Criteria:

* Smoking or any other use of tobacco.
* Taking neuroleptics or benzodiazepines (allowed to take oxazepam ad vesp).
* Neurological-, cardiovascular-, gastrointestinal- or genitourinary disorders of medical importance.
* Glaucoma or history of possibly raised intraocular pressure.
* Impaired liver- or kidney function.
* Hypersensitivity to Scopolamine or any component in the formulation.
* Any indication of drug, alcohol or medicine abuse.
* Participation in another investigational study at the same time.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2004-04; Primary Completion 2004-10 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Changes in EEG as a result of scopolamine administration | 1 hr after scopolamine administration
  The EEG is recorded before, during and after scopolamine administration in order to monitor the effects scopolamine has on the brain as measured by EEG.

CONTACTS AND LOCATIONS:
Overall Officials: Jón Snædal, MD, Principal Investigator — Landspitali University Hospital

REFERENCES:
- [Background] Gudmundsson S, Runarsson TP, Sigurdsson S, Eiriksdottir G, Johnsen K. Reliability of quantitative EEG features. Clin Neurophysiol. 2007 Oct;118(10):2162-71. doi: 10.1016/j.clinph.2007.06.018. Epub 2007 Aug 31. PMID 17765604
- [Result] Snaedal J, Johannesson GH, Gudmundsson TE, Gudmundsson S, Pajdak TH, Johnsen K. The use of EEG in Alzheimer's disease, with and without scopolamine - a pilot study. Clin Neurophysiol. 2010 Jun;121(6):836-41. doi: 10.1016/j.clinph.2010.01.008. Epub 2010 Feb 12. PMID 20153691